CLINICAL TRIAL: NCT02641028
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Design Study of CERC-501 in a Human Laboratory Model of Smoking Behavior
Brief Title: A Study in a Human Laboratory Model of Smoking Behavior
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Clin501-201
Record Dates: First submitted 2015-12-15; First posted 2015-12-29 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Aticaprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CERC-501 (Experimental): Administered orally once daily, 15mg daily, 8 days.
  Interventions: Drug: CERC-501
- Placebo (Placebo Comparator): Administered orally daily, 8 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CERC-501 — CERC-501
  Arms: CERC-501
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Crossover Design Study of CERC-501 in a Human Laboratory Model of Smoking Behavior.

DETAILED DESCRIPTION:
The study will be performed in subjects who are heavy cigarette smokers currently not seeking treatment for tobacco use disorder.

The study is a crossover design study (within-subject analysis), which allows for subjects to be their own control.

Each period of the crossover consists of a 7-day out-patient treatment period followed by a single in-patient testing day on Day 8. Subjects will participate in a laboratory session following the McKee Smoking Lapse Test and be discharged from the clinic to undergo a 7 day washout period followed by the second period of the crossover design and a 7-day follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent and agrees to complete required clinic visits
2. Male or female 21 to 60 years of age inclusive
3. Body mass index (BMI) 18.5 to 40 kg/m2 inclusive
4. Heavy Smokers
5. Currently not seeking smoking cessation therapy
6. In otherwise good general health without any unstable medical conditions (as determined by medical history, medication history, physical examination, 12-lead ECG, vital signs, and clinical laboratory testing)
7. Able to read, write, and speak in English
8. Females must be either:

   * Post-menopausal (amenorrhea for at least 12 consecutive months), surgically sterile -or-
   * Women of childbearing potential (WOCBP) must meet the criteria below:

     * Uses an acceptable double-barrier method of contraception as determined by the Investigator -and-
     * Is not lactating, has a negative serum beta human chorionic gonadotropin pregnancy test at screening and a negative urine pregnancy test prior to dosing on Days 1 and 8 of each treatment period.
9. Male subjects must agree to use a condom if partner is of childbearing potential

Exclusion Criteria:

Subjects meeting the following criteria are not eligible for the study:

1. Any substance use disorder other than nicotine or caffeine as assessed by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) substance use disorder checklist in addition to the Mini-International Neuropsychiatric Interview (MINI) (to capture both DSM-V substance use disorder diagnoses)
2. Current neurological conditions that interfere with study conduct, assessment or treatment in any significant fashion
3. Any lifetime history of bipolar I, II; schizophrenia or any other psychotic disorders; personality disorders, impulse control disorders as assessed by the MINI
4. Current psychiatric conditions that interfere with study conduct, assessment or treatment in any significant fashion, such as major depressive disorder (MDD), eating disorders, post-traumatic stress disorder, etc., without permission of the medical monitor
5. Recent active or past history of gastric disease such as peptic ulcer disease, gastritis, upper gastrointestinal bleeding, or any gastrointestinal malignancy or precancerous condition
6. Active, comorbid disease that might limit the ability of the subject to participate in the study as determined by the Investigator (i.e., poorly controlled diabetes mellitus, congestive heart failure, etc.)
7. Clinically significant clinical laboratory test taken during screening, without permission of the Medical Monitor
8. Elevated AST or ALT ≥ 2 times the upper limit of normal (ULN)
9. Human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C positive as determined by serology testing at Screening
10. History of severe allergies or multiple adverse drug reactions
11. Known hypersensitivity to CERC-501
12. Current use of a proton pump inhibitor or histamine 2 blocker without permission of the Medical Monitor
13. Use of any investigational medication within 2 months prior to the start of this study or scheduled to receive an investigational drug other than the study drug during the course of this study

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2016-09-13 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Latency | 50 min
  Latency (in minutes and seconds) to time of first cigarette smoked during the delay period
Number of Cigarettes smoked | 60 min
  Number of cigarettes smoked during the self administration period

SECONDARY OUTCOMES:
Tobacco Craving | Up to 4 days ( 2 each period)
  Tobacco craving assessed by the Tiffany Questionnaire of Smoking Urges-Brief (QSU-Brief) prior to tobacco withdrawal (Day 7 of each Period) and prior to reinstatement of tobacco (Day 8 of each period)
Mood Scores | Up to 4 days ( 2 each period)
  Mood Scores (Circumplex) prior to tobacco withdrawal (Day 7 of each Period) and prior to reinstatement of tobacco (Day 8 of each period)
Nicotine Withdrawal | Up to 4 days ( 2 each period)
  Nicotine withdrawal scores will be assessed by the Minnesota Nicotine Withdrawal Scale (MNWS) prior to tobacco withdrawal (Day 7 of each Period) and prior to reinstatement of tobacco (Day 8 of each period)
Anxiety Scores | Up to 4 days ( 2 each period)
  Anxiety Scores will be assessed by the Clinically Useful Depression Outcome Scale Modified for Anxious distress (CUDOS-A) prior to tobacco withdrawal (Day 7 of each Period) and prior to reinstatement of tobacco (Day 8 of each period)
Subject Feeling | Up to 4 days ( 2 each period)
  Subject feelings of positive and negative effect of tobacco as assessed by the Modified Cigarette Evaluation Questionnaire (mCEQ) prior to tobacco withdrawal (Day 7 of each Period) and prior to reinstatement of tobacco (Day 8 of each period)
Electronic Diary | up to 51 days
  Daily Smoking Diary for out-patient periods

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Marcus, MD, Study Director — Avalo Therapeutics, Inc.
Locations (3):
- United States (3):
  - Vince and Associates, Overland Park, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No